CLINICAL TRIAL: NCT02403869
Title: Study of Quality of Life in Patients With Metastatic Breast Cancer Treated With Second-line Monochemotherapy
Brief Title: Quality of Life in Metastatic Breast Cancer (MBC) Patients in Second Line Monochemotherapy
Acronym: DD-CMM
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-CMM-2013-01
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Breast Neoplasms
Keywords: Metastatic breast cancer; Monotherapy; chemotherapy; second line; treatment; Her 2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: MBC patients starting treatment with monochemotherapy for second line of quimiotherapy treatment for metastatic disease

SUMMARY:
Post-authorization, prospective follow-up, multi-centre, national study to estimate definitive deterioration in the quality of life in patients with metastatic breast cancer treated with second-line monochemotherapy.

DETAILED DESCRIPTION:
Post-authorization, prospective, multi-centre study in Metastatic Breast Cancer patients treated with second-line monochemotherapy.

A total of 200 patients are expected to be recruited from 32 Spanish sites.

In this study the results perceived by patients will be compiled to assess overall Quality of Life (QoL) in MBC patients treated with second-line monochemotherapy, using the EORTC QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) and its modules EORTC QLQ-BR23 (EORTC Breast Cancer specific) and EORTC QLQ-CIPN20 (EORTC Chemotherapy-Induced Peripheral Neuropathy).

Patients will be evaluated at the time of acceptance to participate in the study after signing the informed consent and will be tracked every three months during treatment with second-line monochemotherapy, coinciding with routine assessments within normal clinical practice. When the patient completes treatment with second-line chemotherapy he/she will enter the post-treatment period, with follow-up at six and 12 months after completion of treatment. Also, patients will be followed to assess survival until the end of the study (30 months after enrolment of the last patient in the study). Follow-up time has been established based on the median survival of patients with MBC

ELIGIBILITY:
Inclusion Criteria:

* Patients who give their written informed consent.
* Patients with metastatic breast cancer who start treatment with second-line monochemotherapy.
* Patients of both sexes, at least 18 years of age and of any race.
* Patients with life expectancy longer than or equal to 12 weeks.
* Patients with histological or cytological diagnosis of Her-2/neu negative breast adenocarcinoma.
* Patients with ability enough to understand the questionnaires.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients who have been treated with chemotherapy in the last three weeks
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MBC patients, older than or equal to 18 years of age, on second line of treatment with chemotherapy regimens in monotherapy and Her-2/neu-negative status
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Definitive deterioration at 6 months | 6 months
  Proportion of patients with definitive deterioration at six months after initiation of second-line mono-chemotherapy for MBC

SECONDARY OUTCOMES:
Definitive deterioration at 3 months | 3 Months
  Description Proportion of patients with definitive deterioration at 3 months after the start of the second-line mono-chemotherapy and at the time of disease progression or completion of treatment for other reasons
Definitive deterioration at 9 months | 9 Months
  Proportion of patients with definitive deterioration at 9 months after the start of the second-line mono-chemotherapy and at the time of disease progression or completion of treatment for other reasons
Definitive deterioration at 12 months | 12 Months
  Proportion of patients with definitive deterioration at 12 months after the start of the second-line mono-chemotherapy and at the time of disease progression or completion of treatment for other reasons
Time to Definitive deterioration (TTDD) | Up to 42 months
  Estimated median TTDD using the actuarial method
Overall survival | Up to 42 months
  Estimated overall survival using the Kaplan-Meier method
TTDD as a prognostic factor | Up to 42 months
  Determine if TTDD is an independent prognostic factor for overall survival using Cox regression.
Quality of life | Up to 42 months
  Comparison of the mean score of the scales of the EORTC QLQ-C30, EORTC QLQ-BR23 and between patients ≥70 years and <70 years at baseline, every 3 months approximately and at the time of disease progression or completion of treatment for other reasons
Quality of life every 3 months | Up to 42 months
  Score in the scales of the EORTC QLQ-C30 and EORTC QLQ-BR23 questionnaires at baseline, every 3 months approximately and at the time of disease progression or completion of treatment for other reasons.
Chemotherapy-induced peripheral neuropathy | Up to 42 months
  Incidence, management and duration of chemotherapy-induced peripheral neuropathy at baseline, every 3 months approximately up to disease progression and at 6 and 12 months after completion of second-line chemotherapy
Chemotherapy-induced peripheral neuropathy in the EORTC QLQ-CIPN20 | Up to 42 months
  Assess the effect of chemotherapy-induced peripheral neuropathy in the EORTC QLQ-CIPN20 quality of life questionnaire at baseline, every 3 months approximately up to disease progression or completion of treatment for other reasons and at 6 and 12 months after completion of second-line chemotherapy
Definitive deterioration | Up to 42 months
  Comparison of the proportion of patients with definitive deterioration at every 3 months approximately up to disease progression or completion of treatment for other reasons in patients with ECOG 0-1 and ECOG 2-3, using the chi-squared test.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- Spain (29):
  - Hospital Juan Ramón Jiménez, Huelva, Andalusia
  - Hospital Virgen de Valme, Seville, Andalusia
  - Hospital Virgen del Rocío, Seville, Andalusia
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Son Espases, Palma Mallorca, Balearic Islands
  - Hospital Universitario Canarias, La Laguna, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Burgos, Burgos, Castille and León
  - Complejo Hospitalario de León, León, Castille and León
  - Hospital Bierzo, León, Castille and León
  - Hospital Universitario Salamanca, Salamanca, Castille and León
  - Hospital Virgen de la Salud. Toledo, Toledo, Castille-La Mancha
  - Centro Médico Teknon, Barcelona, Catalonia
  - Hospital Clinic Barcelona, Barcelona, Catalonia
  - Hospital Universitario San Joan de Reus, Reus, Tarragona, Catalonia
  - Corporación Sanitaria Parc Taulí- Sabadell, Sabadell, Catalonia
  - H. Infanta Cristina de Badajoz, Badajoz, Extremadura
  - H. San Pedro de Alcántara, Cáceres, Extremadura
  - Complejo Hospitalario de Ourense, Ourense, Galicia
  - Complejo Hospitalario de Pontevedra-Montecelo, Pontevedra, Galicia
  - Complejo Hospitalario Universitario de Santiago Compostela, Santiago de Compostela, Galicia
  - Complejo Hospitalario de Vigo, Vigo, Galicia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Elche, Elche, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Infanta Sofía, Madrid